CLINICAL TRIAL: NCT05919095
Title: A Single-arm, Multicenter, Phase II Clinical Study of the Efficacy and Safety of Carrilizumab Combinated With Gemcitabine and Oxaliplatin (GEMOX) as a Preoperative Translational Therapy for Unresectable Gallbladder Cancer
Brief Title: A Clinical Study of a Preoperative Translational Therapy for Unresectable Gallbladder Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2022-516-02
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Unresectable Gallbladder Cancer
Keywords: PD-1；GEMOX；Unresectable gallbladder cancer.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carrilizumab plus GEMOX (Experimental): Carrilizumab combinated With gemcitabine and oxaliplatin (GEMOX)
  Interventions: Drug: Carrilizumab plus GEMOX

INTERVENTIONS:
Drug: Carrilizumab plus GEMOX — PD-1 antibody，200mg，D1，intravenous infusion, the administration time is 60 (+15) minutes.
  GEMOX chemotherapy : gemcitabine 1000mg/m2,D1，D8；oxaliplatin 100mg/m2,D1intravenous infusion.Three weeks is a course of treatment.

SUMMARY:
This is an open-label,multicenter ,non-randomized,single arm exploratory study. The objective of this study is to evaluate the efficacy and safety of PD-1 antibody plus GEMOX as preoperative translational therapy for unresectable gallbladder cancer.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the efficacy and safety of carrilizumab in combination with gemcitabine and oxaliplatin (GEMOX) as a preoperative conversion therapy for unresectable gallbladder cancer. Patients with unresectable gallbladder cancer were enrolled to receive gemcitabine 1000 mg/m2 D1, D8 + oxaliplatin 100 mg/m2, D1 + carrilizumab 200 mg, D1, in 21-day cycles for 6-8 cycles, with changes in serum tumor parameters assessed at each course and abdominal CTA performed every two courses.The above treatment was terminated if the CT evaluation revealed disease progression, and the investigator could adjust the treatment regimen according to the guideline. The primary outcome measure of this study is the tumor radical resection rate; secondary outcome measure are objective response rate, disease control rate, progression-free survival, and overall survival. The safety indicators are the incidence and severity of adverse events (AE) and serious adverse events (SAE) according to NCI-CTCAEv5.0 criteria. Thirty-seven cases are expected to be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must sign an informed consent form;
2. Age 18-75 years old, both male and female;
3. ECOG performance status score (PS score) 0 or 1 point;
4. Child-Pugh score A period;
5. Patients with advanced or recurrent metastatic gallbladder cancer who are not suitable for radical surgery (R0), or non-radical surgery (R1), or palliative surgery, as confirmed by pathological histology or cytology.
6. Have not received any systemic treatment within 6 months;
7. The functional indicators of important organs meet the following requirements (1)Neutrophils≥1.5*109/L; platelets≥100*109/L; hemoglobin≥9g/dl; serum albumin≥3g/dl; (2)Thyroid-stimulating hormone (TSH) ≤ 2 times the upper limit of normal, and T3 and T4 are in the normal range; (3)Bilirubin ≤ 1.5 times the upper limit of normal; ALT and AST ≤ 3 times the upper limit of normal; (4)Serum creatinine ≤ 1.5 times the upper limit of normal, and creatinine clearance ≥ 60ml/min (calculated by Cockcroft-Gault formula);
8. The subject has at least 1 measurable lesion (according to RECIST1.1);
9. For women who are not breastfeeding or pregnant, use contraception during treatment or 12 months after the end of treatment.

Exclusion Criteria:

1. Past or simultaneous suffering from other malignant tumors, except for fully treated non-melanoma skin cancer, cervical carcinoma in situ, and thyroid papillary carcinoma;
2. Have used gemcitabine-based chemotherapy or have used PD-1 monoclonal antibody or PD-L1 monoclonal antibody treatment within 6 months;
3. Severe cardiopulmonary and renal dysfunction;
4. Hypertension that is difficult to control with drugs (systolic blood pressure (BP) ≥140 mmHg and/or diastolic blood pressure ≥90mmHg) (based on the average of ≥3 BP readings obtained by ≥2 measurements);
5. Abnormal coagulation function (PT>14s), have bleeding tendency or are receiving thrombolysis or anticoagulation therapy;
6. After antiviral treatment, HBV DNA>2000 copies/ml, HCV RNA>1000;
7. A history of esophageal and gastric varices, significant clinically significant bleeding symptoms or a clear tendency to appear within 3 months before enrollment;
8. Active infections requiring systemic treatment; patients with active tuberculosis infection within 1 year before enrollment; a history of active tuberculosis infection more than 1 year before enrollment, and no formal anti-tuberculosis treatment or tuberculosis Still in the active period;
9. Human immunodeficiency virus (HIV, HIV1/2 antibody) positive;
10. A history of psychotropic drug abuse, alcohol or drug abuse;
11. Known to have a history of severe allergies to any monoclonal antibodies, platinum drugs, or gemcitabine;
12. Other factors judged by the investigator may affect the safety of the subjects or the compliance of the trial. Such as serious diseases (including mental illness) that require combined treatment, serious laboratory abnormalities, or other family or social factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Radical resection rate | 6 months
  The proportion of patients whose tumors converted to a surgically resectable state and achieved radical resection within 8 courses of medication in all patients enrolled.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 6 months
  Complete response (CR) and partial response (PR), at 6 months by RECIST v.1.1
Disease control rate(DCR) | 6 months
  Complete response (CR) ,partial response (PR) and stable disease, SD, at 6 months by RECIST v.1.1
Progression-free survival (PFS) | 6 months
  The time from first drug administration to the first documented disease progression according to RECIST version 1.1 or to death from any cause, whichever occurred first.
Overall survival(OS) | 6 months
  The time from first drug administration to death from any cause.
The incidence of treatment-related adverse event | 6 months
  Percentage of participants who experienced treatment-related adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Rui Zhang, PhD, Principal Investigator — Department of Biliary and Pancreatic Surgery, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baiu I, Visser B. Gallbladder Cancer. JAMA. 2018 Sep 25;320(12):1294. doi: 10.1001/jama.2018.11815. No abstract available. PMID 30264121
- [Background] Lamarca A, Palmer DH, Wasan HS, Ross PJ, Ma YT, Arora A, Falk S, Gillmore R, Wadsley J, Patel K, Anthoney A, Maraveyas A, Iveson T, Waters JS, Hobbs C, Barber S, Ryder WD, Ramage J, Davies LM, Bridgewater JA, Valle JW; Advanced Biliary Cancer Working Group. Second-line FOLFOX chemotherapy versus active symptom control for advanced biliary tract cancer (ABC-06): a phase 3, open-label, randomised, controlled trial. Lancet Oncol. 2021 May;22(5):690-701. doi: 10.1016/S1470-2045(21)00027-9. Epub 2021 Mar 30. PMID 33798493
- [Background] Song X, Hu Y, Li Y, Shao R, Liu F, Liu Y. Overview of current targeted therapy in gallbladder cancer. Signal Transduct Target Ther. 2020 Oct 7;5(1):230. doi: 10.1038/s41392-020-00324-2. PMID 33028805
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Morizane C, Okusaka T, Mizusawa J, Katayama H, Ueno M, Ikeda M, Ozaka M, Okano N, Sugimori K, Fukutomi A, Hara H, Mizuno N, Yanagimoto H, Wada K, Tobimatsu K, Yane K, Nakamori S, Yamaguchi H, Asagi A, Yukisawa S, Kojima Y, Kawabe K, Kawamoto Y, Sugimoto R, Iwai T, Nakamura K, Miyakawa H, Yamashita T, Hosokawa A, Ioka T, Kato N, Shioji K, Shimizu K, Nakagohri T, Kamata K, Ishii H, Furuse J; members of the Hepatobiliary and Pancreatic Oncology Group of the Japan Clinical Oncology Group (JCOG-HBPOG). Combination gemcitabine plus S-1 versus gemcitabine plus cisplatin for advanced/recurrent biliary tract cancer: the FUGA-BT (JCOG1113) randomized phase III clinical trial. Ann Oncol. 2019 Dec 1;30(12):1950-1958. doi: 10.1093/annonc/mdz402. PMID 31566666
- [Background] Chen X, Wu X, Wu H, Gu Y, Shao Y, Shao Q, Zhu F, Li X, Qian X, Hu J, Zhao F, Mao W, Sun J, Wang J, Han G, Li C, Xia Y, Seesaha PK, Zhu D, Li H, Zhang J, Wang G, Wang X, Li X, Shu Y. Camrelizumab plus gemcitabine and oxaliplatin (GEMOX) in patients with advanced biliary tract cancer: a single-arm, open-label, phase II trial. J Immunother Cancer. 2020 Nov;8(2):e001240. doi: 10.1136/jitc-2020-001240. PMID 33172881
- [Background] Creasy JM, Goldman DA, Dudeja V, Lowery MA, Cercek A, Balachandran VP, Allen PJ, DeMatteo RP, Kingham PT, D'Angelica MI, Jarnagin WR. Systemic Chemotherapy Combined with Resection for Locally Advanced Gallbladder Carcinoma: Surgical and Survival Outcomes. J Am Coll Surg. 2017 May;224(5):906-916. doi: 10.1016/j.jamcollsurg.2016.12.058. Epub 2017 Feb 13. PMID 28216422
- [Background] Chaudhari VA, Ostwal V, Patkar S, Sahu A, Toshniwal A, Ramaswamy A, Shetty NS, Shrikhande SV, Goel M. Outcome of neoadjuvant chemotherapy in "locally advanced/borderline resectable" gallbladder cancer: the need to define indications. HPB (Oxford). 2018 Sep;20(9):841-847. doi: 10.1016/j.hpb.2018.03.008. Epub 2018 Apr 26. PMID 29706425
- [Background] Kato A, Shimizu H, Ohtsuka M, Yoshitomi H, Furukawa K, Takayashiki T, Nakadai E, Kishimoto T, Nakatani Y, Yoshidome H, Miyazaki M. Downsizing Chemotherapy for Initially Unresectable Locally Advanced Biliary Tract Cancer Patients Treated with Gemcitabine Plus Cisplatin Combination Therapy Followed by Radical Surgery. Ann Surg Oncol. 2015 Dec;22 Suppl 3:S1093-9. doi: 10.1245/s10434-015-4768-9. Epub 2015 Aug 4. PMID 26240009
- [Background] Liu QQ, Lin HM, Han HW, Yang CN, Liu C, Zhang R. Complete Response to Combined Chemotherapy and Anti-PD-1 Therapy for Recurrent Gallbladder Carcinosarcoma: A Case Report and Literature Review. Front Oncol. 2022 Mar 14;12:803454. doi: 10.3389/fonc.2022.803454. eCollection 2022. PMID 35372010